CLINICAL TRIAL: NCT05835440
Title: Improving Wrist Injury Pathways (I-WIP): a Qualitative Study
Brief Title: Improving Wrist Injury Pathways (I-WIP) Study
Acronym: I-WIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: AO Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 321650
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Scaphoid Fracture; Wrist Injuries
MeSH Terms: conditions — Wrist Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- staff stakeholders: The potential stakeholders are a diverse population and will include managers, emergency department clinicians and practitioners, radiologists, radiographers, administrative staff and surgeons. A maximum total of 4 staff stakeholder interviews shall be undertaken.
  Interventions: Other: no intervention
- patient participants: The patient population are adults who have sustained a traumatic wrist injury with normal X-rays and have been treated by NHS services.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — interviews

SUMMARY:
Wrist injuries represent a considerable problem for both patients and the NHS. Around 70,000 patients per year in the UK attend hospitals with serious wrist pain after an injury, only to find that their x-ray is considered to be 'normal'. The National Institute of Care and Health Excellence (NICE) advises that these patients should be given MRI (magnetic resonance imaging) scans early on, within 2 weeks. Early MRI gives patients the best care, by picking up the serious injuries requiring early treatment and by helping reassure those without serious injuries to get back to activities quickly. This saves the NHS staff time and money by reducing unnecessary clinic attendances. Although these benefits from early use of MRI scans, and the NICE guidance, are clear, it is know from our recent national (UK) survey that only 11 of the 87 UK hospitals that we surveyed used MRI scans for these patients.

The gap between what the best evidence suggests and what happens in clinical practice is a complex issue that requires further investigation. To develop a complex intervention to address this problem,a better understanding of the reasons why hospital services are currently unable to adopt the NICE guidance is needed. Clinical interventions in surgery exist on a spectrum from simple, such as closing a wound with stitches, to the complicated (carrying out a joint replacement for a neck of femur fracture) to complex (improving trauma theatre efficiency). The latter, more complex variety, are characterised by the 1) number of components in the intervention, 2) the range of behaviours targeted 3) the range and different levels of target recipients, 4) the expertise and skills required by those delivering and receiving the intervention 5) and or by the level of flexibility permitted in the intervention delivery. In 2000, the UK Medical Research Council (MRC) established guidance for developing and evaluating complex interventions to improve the delivery of health care services. An important stage in developing complex interventions and improving care is to fully understand current pathways and the context of care. This qualitative study aims to develop a better understanding of wrist injury pathways, and their context, in the NHS. We aim to (1) understand the barriers to early MRI for painful wrists and (2) understand what is important to patients when being treated with a wrist injury.

DETAILED DESCRIPTION:
Around 70,000 patients per year in the UK attend hospitals with serious wrist pain after an injury, which although painful on examination, look 'normal' on x-ray. The National Institute of Care and Health Excellence (NICE) advises that this large group of patients who have pain, but normal x-rays, should be given MRI (magnetic resonance imaging) scans early on. Early MRI gives patients the best care, by picking up the serious injuries requiring early treatment and by enabling those without serious injuries to get back to activities quickly after being reassured and potentially saves NHS resource by reducing unnecessary clinic attendances(1). Although these benefits from early use of MRI scans, and the NICE guidance, are clear, it is known from our recent national (UK) survey that MRI scans are underused around the country. Only 13% (11 of 87) of centres currently use MRI directly for patients(2).

There are multiple, often complicated reasons, for centres not being able to follow the NICE guidance, however when they do use MRI scans early on, it makes patients better faster, and saves the NHS money(3). This implementation gap between what best evidence recommends and what happens in clinical practice is a complex issue that requires further investigation. To develop an effective complex intervention to address this problem, a far better understanding of the reasons underlying this failure to implement NICE guidance is needed. In 2000, the UK Medical Research Council (MRC) established guidance for developing and evaluating complex interventions to improve the delivery of health care services(4).This guidance advises that six core elements are considered when developing a complex intervention:

1. How does the intervention interact with its context?
2. What is the underpinning programme theory?
3. How can diverse stakeholder perspectives be included in the research?
4. What are the key uncertainties?
5. How can the intervention be refined?
6. Do the effects of the intervention justify its cost?

A vital early task in ensuring evidence-based treatment of wrist injuries is to develop a theoretical understanding of the drivers (or root causes) of the problem. To do this, we need to draw on existing evidence and theory from similar contexts, and verify our initial assumptions through primary research, for example interviews with stakeholders and the detailed mapping of care pathways. In this case, the relevant stakeholders are a highly diverse group including commissioners, managers, ED staff (including doctors, paramedics, nurses and other allied health professionals), administrative staff, radiologists, radiographers and surgical staff (including surgeons, nurses, physiotherapists and other allied health professionals).

It will be important to consider the potential barriers and facilitators to complex interventions in orthopaedic surgery. The Donabedian model of quality assessment is useful here(5). This model proposes that any given outcome (in this case early MRI of the wrist) is the product of (a) process factors (the way care is organised or delivered) and (b) structural factors (the physical capacity of the service to deliver the target outcome). Our exploratory work has demonstrated deeply entrenched negative views regarding the value of early MRI which are likely to be a barrier to change in some centres. MRI capacity may be a significant barrier to implementation. Process barriers might include inefficient use of existing MRI capacity, which would be amenable to pathway implementation to streamline and improve efficiency. Conversely structural problems, such as insufficient capacity despite optimising MRI efficiency may require the purchase of more scanners and recruitment of more staff. Structural problems are harder to influence with behaviour change interventions and generally need a different approach e.g., business case or funding (6).

This qualitative study aims to develop a better understanding of wrist injury pathways in the NHS.

Although it is not expected for harm to come to participants from the interview, qualitative interviews encourage people to talk about a range of subjects that can be upsetting. Our experience has shown us that talking can be a positive experience for many people. The participants will be interviewed by a trained NHS clinician who will direct any patients who experience worrying distress to the appropriate healthcare professional or encourage the person to speak to their GP. The interviewer will also structure the interview with a 'cool off' time at the end.

ELIGIBILITY:
Inclusion Criteria

- All participants are willing and able to give informed consent for participation in the study (including audio recording of interview). Where possible we shall use translation services to enable those who might not adequately understand various forms of information to take part

For staff stakeholders (NHS staff) - Any staff member involved in regular delivery or management of Wrist Injury Pathways (e.g. manager, nurse practitioner, physiotherapist, surgeon, administrative staff, radiologist, radiographer, emergency department clinician). This staff member must be deemed to be integral in the day to day running and/or overall management of the pathway.

For patients:

* Male or female aged over 18 years of age
* Being treated for a traumatic wrist injury with a normal initial X-ray

Exclusion Criteria

- Learning difficulty

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For aim 1, the staff stakeholders (NHS staff) shall be identified using snowballing sampling starting with the local QI project lead and the aim is to undertake up to 40 staff stakeholder interviews (maximum of 4 at each site).
  For aim 2, we will undertake up to 30 patient participant interviews recruited from trauma clinics (3 at each site). As explained above, patient participants shall be sampled purposively to achieve a diversity in terms of gender and age.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Thematic analysis of interview data | 12 months
  thematic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- OUH NHS TRust, Oxford, Oxon, United Kingdom

IPD SHARING:
Plan to Share IPD: No